CLINICAL TRIAL: NCT05234658
Title: Phase II Clinical Trial Evaluating the Safety and Efficacy of a Tissue Engineered Autologous Skin Substitute Reconstructive Surgery for Basal Cell Carcinoma
Brief Title: Study of an Artificial Human Skin Medicine for Patients With Basal Cell Carcinoma Undergoing Reconstructive Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NanoGSkin-CB-2019
Record Dates: First submitted 2021-12-27; First posted 2022-02-10 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PHIT (Experimental): Human artificial skin created by tissue engineering, composed of a sheet of autologous adult differentiated skin keratinocytes and fibroblasts expanded in a biological fibrin-agarose matrix (PHIT).
  Interventions: Biological: PHIT
- PHITAH (Experimental): Human artificial skin created by tissue engineering, composed of a sheet of keratinocytes and differentiated autologous adult skin fibroblasts expanded in a biological fibrin-hyaluronic matrix (PHITAH).
  Interventions: Biological: PHITAH
- Skin Autograft (Active Comparator): Skin autograft.
  Interventions: Biological: Skin Autograft

INTERVENTIONS:
Biological: PHITAH — Tissue Engineered Human Artificial Skin: Fibrin-Hyaluronic Acid
  Arms: PHITAH
Biological: PHIT — Human artificial skin created by tissue engineering: fibrin-agarose
  Arms: PHIT
Biological: Skin Autograft — Skin Autograft
  Arms: Skin Autograft

SUMMARY:
Phase II Clinical Trial Evaluating the Safety and Efficacy of a Tissue Engineered Autologous Skin Substitute Reconstructive Surgery for Basal Cell Carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Patients that give their informed consent for study participation.
2. Adult (18 years of age or older), of any sex and racial origin.
3. Clinical and dermatoscopic diagnosis of basal cell carcinoma with lesions on the scalp, torso or extremities, within a certain size that do not allow for surgical closure by direct suture or flaps. Namely, indication for Mohs surgery.
4. Women with childbearing age or men capable of producing a child, should commmit to use contraceptives of medically proven efficacy.

Exclusion Criteria:

1. Locally advanced basal cell carcinoma with evidence of tissue infiltration.
2. Lesions in the face.
3. Injuries requiring urgent surgical intervention.
4. Infected lesions, necrosis, scarcely vascularized injuries or other complications that may interfere with healing and/or integrity of the graft.
5. Injuries that have received treatment with radiotherapy.
6. Contraindication for Mohs surgery.
7. Known allergies to Biobrane dressing.
8. Pregnant or breastfeeding women.
9. Coexistence of any other pathology that, in the investigator's opinion, could compromise the healing process or interfere with protocol follow-up.
10. Participation in other clinical trials in 3 months previous to inclusion, or in the previous 5 years for trials with advanced therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety of autologous bioengineered skin | Through study completion, an average of 2 year
  Incidence of adverse events related to investigational medicinal products
Efficacy of autologous bioengineered skin | Through study completion, an average of 2 year
  Satisfaction of the graft assessed by doppler ultrasound and study of homeostasis

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital Costa del Sol, Marbella, Málaga
  - Hospital U. Virgen de las Nieves, Granada
  - Hospital U. Virgen de la Victoria, Málaga
  - Hospital U. Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: No